Official Title: Diamox/Aldactone to Increase the URinary Excretion of Sodium: an Investigational Study in Congestive Heart Failure

NCT01973335

Date: August 27, 2015

## 1. Background

Aging of the population and prolongation of the lives of cardiac patients by modern therapeutic innovations have led to an increased incidence of congestive heart failure (CHF).¹ During the last two decades, important progress has been made in the treatment of ambulatory CHF patients with reduced ejection fraction. Renin-angiotensin system blockers, β-blockers, mineralocorticoid receptor antagonists (MRA), ivabradine and cardiac resynchronization therapy have all demonstrated to reduce morbidity and/or mortality in ambulatory CHF patients.²-¹¹ Despite these important advances, many patients are still hospitalized frequently with signs and symptoms of systemic congestion, which is associated with worse outcome.¹¹ Treatment in these cases mainly focuses on symptomatic relief through administration of diuretics, although clear evidence on the optimal agent, dosing schedule, and administration route is lacking.

Coexisting renal dysfunction often complicates decongestive treatment and worsening renal function (WRF), often defined as a 0.3 mg/dL rise in serum creatinine (Cr), is a common finding in this context.<sup>19</sup> However, the prognostic impact of WRF, defined as Cr change is unsure as it might be associated with worse, neutral or even better outcome.<sup>20-22</sup> In contrast, persistent congestion, as a reflection of the inability of the kidneys to preserve sodium homeostasis, has been more consistently associated with higher mortality and more frequent readmissions in CHF.<sup>23</sup> This suggests that achieving a negative sodium balance might be an attractive treatment target in heart failure.

Loop diuretics are by far the most commonly used diuretic agents to achieve a negative sodium balance in acute decompensated heart failure (ADHF). Especially in diuretic-naïve patients, they are often very effective to relief dyspnea and congestive symptoms. However, in the recent Diuretic Optimization Strategies Evaluation (DOSE) trial, no differences in patients' global assessment of symptoms or change in renal function were observed when loop diuretics were administered by bolus as compared with continuous

infusion or at high versus low dose during a hospitalization for ADHF, with high dose therapy currently considered as usual care by most clinicians.24 Importantly, there are several reasons why loop diuretics might be less effective or even harmful in CHF. First, loop diuretics directly stimulate renin production by inhibiting the Na<sup>+</sup>/K<sup>+</sup>/2Cl<sup>-</sup>-cotransporter on the luminal side of the macula densa, which depletes intracellular chloride levels in the macula densa. The consequence is an increased COX-2 and NOS I activity in macula densa cells, leading to paracrine PGE2 and NO secretion.25 Both PGE2 and NO work in concert to stimulate renin release by granulosa cells of the afferent arteriole and further detrimental activation of the renin-angiotensin-aldosterone axis. Second, impaired secretion of loop diuretics in the proximal tubules of CHF patients, especially when there is concomitant renal dysfunction, results in lower concentrations at the place where these agents act – the luminal side of the thick ascending limb of Henle's loop (TAL). Third, increased sodium reabsorption in the proximal tubules might result in less sodium offered to the TAL, especially if glomerular filtration is concomitantly impaired, hampering the efficacy of loop diuretics. As a result, physicians often use combination therapies of different acting diuretic agents in order to increase the overall diuretic effect.

From a pathophysiological point of view, targeting sodium reabsorption in the proximal tubules has several potential benefits in CHF. First, it is the place where most sodium is reabsorbed, especially in ADHF. Second, greater delivery of chloride to macula densa cells will decrease renin production, ceasing neurohumoral activation. Third, endogenous natriuretic peptides (acting in the distal nephron) will possibly regain their effects. The carbonic anhydrase inhibitor acetazolamide (Diamox®), which is approved for the treatment of mountain sickness and is used to increase the diuretic efficacy of loop diuretics in patients with therapy-refractory congestion, inhibits sodium reabsorption in the proximal tubules. Remarkably, in a small study of 9 patients with advanced CHF and diuretic resistance, therapy with acetazolamide was able to elicit potent diuresis.<sup>26</sup> Despite this

promising case series and the pathophysiological rationale for inhibition of proximal sodium reabsorption in ADHF, acetazolamide is now a largely forgotten diuretic.

MRA have an established role in the treatment of chronic CHF.<sup>11, 12</sup> However there are remarkable few data on their use in patients who present with ADHF. Nevertheless, in this context with frequent use of potassium wasting diuretics, they might be of particular interest to prevent occurrence of hypokalemia, which has been associated with a worse prognosis.<sup>27</sup> Moreover, by inhibiting distal tubular sodium reabsorption and counteracting aldosterone breakthrough, MRA might improve the natriuretic efficiency of loop diuretics.

## 2. Study Hypotheses

- Combination therapy with acetazolamide improves loop diuretic efficacy to induce natriuresis in ADHF patients, allowing for a lower dose of the latter medication and potentially less adverse events such as worsening renal function.
- Combination therapy with acetazolamide and low-dose loop diuretics leads to less pronounced neurohumoral activation compared to treatment with high-dose loop diuretics in ADHF patients.
- Upfront therapy with MRA is safe in patients presenting with ADHF and lowers the incidence of hypokalemia and the need for potassium supplementation, without causing a higher incidence of hyperkalemia.
- Combination diuretic therapy with acetazolamide and/or upfront spironolactone will lead to improved clinical outcome (less heart failure rehospitalizations and lower all-cause mortality).

# 3. Study Protocol

#### 3.1. Study design

Randomized clinical trial with factorial 2x2 design, 2 treatment arms, and 4 groups (n=20 each):

- Arm 1: <u>Acetazolamide + low-dose loop diuretics</u> versus <u>high-dose loop diuretics</u>
   (=standard of care)
  - → Triple blinded to treatment allocation (patient, treating physician and investigator blinded)
- Arm 2: Upfront versus discharge spironolactone
  - → Treating physician and investigator blinded to treatment allocation. Patient not blinded to treatment allocation because no matching placebo will be provided due to logistic constraints.

Consecutive patients, presenting with ADHF at different Belgian hospitals will be screened by staff members, cardiology fellows, a study nurse and the cardiology Ph.D. fellows. All those people will be able to login via the website <a href="www.hartcentrumlimburg.be">www.hartcentrumlimburg.be</a>, where they can print the case report form and informed consent of the study and will receive the randomization number by a computer algorithm with blocks of 4.

## 3.2. Study population

#### 3.2.1. Inclusion criteria

- Older than 18 years of age and able to give informed consent
- Clinical diagnosis of ADHF within the previous 8 h
- At least two clinical signs of congestion (e.g. edema, ascites, jugular venous distension or pulmonary vascular congestion on chest radiography)
- Maintenance therapy with oral loop diuretics at a dose of at least 1 mg bumetanide or an equivalent dose for at least 1 month before hospital admission
   Conversion: 1 mg bumetanide = 40 mg furosemide = 20 mg torsemide
- Plasma NT-proBNP >1,000 pg/mL
- Left ventricular ejection fraction <50% (on examination ≤3 months)</li>
- One out of three of the following criteria:
  - Serum sodium <136 meg/L</li>

- Urea/creatinine ratio >50
- WRF defined as a >0.3 mg/dL increase in Cr compared to a previous value within 3 months before admission

#### 3.2.2. Exclusion criteria

- History of a cardiac transplantation and/or ventricular assist device
- Concurrent diagnosis of an acute coronary syndrome defined as typical chest pain and/or electrocardiographic changes in addition to a troponine rise >99<sup>th</sup> percentile
- Systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg at the moment of admission
- Use of intravenous inotropes, vasopressors or nitroprusside at any time point during the study
- A baseline estimated glomerular filtration rate <15 mL/min/1.73m² according to the</li>
   Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
- Use of renal replacement therapy or ultrafiltration before study inclusion
- Treatment with acetazolamide during the previous month
- Treatment with ≥2 mg bumetanide or an equivalent dose of loop diuretics during the index hospitalization before randomization
- Use of diuretics or MRA not specified by the protocol
- Exposure to nephrotoxic agents (i.e. contrast dye) anticipated within 3 days

## 3.3. Interventions (See Addendum 1 for therapy schedules)

## 3.3.1. Arm 1, control group: High-dose loop diuretics

- At the moment of randomization the patient receives an intravenous bolus of loop diuretics at a dose equal to the double of his normal daily oral dose (e.g. a patient who takes 1x1 mg burnetanide will receive 2x1x1 mg = 2mg; or a patient who takes 2x1 mg burnetanide will receive 2x2x1 mg = 4mg).
- The next three days, the patient will receive the same dose equally divided between two administrations at 10u00 and 16u00 provided that the treating physician has concluded during the morning rounds that the patient is still volume overloaded.
- If diuresis since administration of the previous dose of loop diuretics is <1,500 mL and the patient is still volume overload, subsequent bolus doses are doubled.
- If after doubling of the dose, the patient is considered therapy-refractory. The treating
  physician is recommended to add chlorthalidone 50mg once daily and consider
  ultrafiltration or renal replacement therapy after which results of the patient will be
  censored.
- Switch to treatment at the discretion of the treating physician if any of the following criteria is fulfilled
  - After 3 days
  - The patient had no longer clinical signs or symptoms of congestion
  - Doubling of the serum creatinine value

## 3.3.2. Arm 1, treatment group: Acetazolamide + low-dose loop diuretics

- At the moment of randomization, the patient receives 500 mg of intravenous acetazolamide and 2 mg of intravenous bumetanide in bolus.
- The next three days, the patient will receive 250 mg of intravenous acetazolamide and 1 mg of intravenous burnetanide in bolus at 10u00 provided that the treating physician has concluded during the morning rounds that the patient is still volume overloaded.

- If diuresis since administration of the previous dose of loop diuretics is <1,500 mL and the patient is still volume overloaded, the patient continues to receive 500 mg of acetazolamide and 2 mg of burnetanide.
- If after doubling of the dose, the patient is considered therapy-refractory. The treating
  physician is recommended to add chlorthalidone 50mg once daily and consider
  ultrafiltration or renal replacement therapy after which results of the patient will be
  censored.
- Switch to treatment at the discretion of the treating physician if any of the following criteria is fulfilled
  - After 3 days
  - The patient had no longer clinical signs or symptoms of congestion
  - Doubling of the serum creatinine value

### 3.3.3. Arm 2, control group: Discharge spironolactone

This group will receive no active treatment. No placebo will be provided either due to logistic constraints. As instructed by the guidelines, addition of a MRA to maintenance therapy will be recommended upon discharge from the hospital.

### 3.3.4. Arm 2, treatment group: Upfront spironolactone

This group will receive oral spironolactone 25 mg immediately after randomization and subsequently each day in the morning (10u00) provided serum potassium levels are <5.0 mmol/L. If no contraindications emerge during hospitalization, spironolactone will be added to the maintenance therapy of the patient upon hospital discharge.

#### 3.3.5. All groups

All groups will receive the same maintenance intravenous therapy with 500 mL Glucose 5% and 3g MgSO4 administered over a 24enin-angiotensin system blockers and  $\beta$ -blockers) will be continued at the discretion of the treating physician, but they are recommended to keep maintenance dosages unchanged.

#### 3.4. Collected data

- Baseline at the moment of randomization
  - Demographics, medical history, current medical therapy, baseline body weight, blood pressure, heart rhythm (sinus or not), heart rate,
     Visual-analogue scale (VAS) score for dyspnea and 4-point Likert scale for edema will be assessed upon study inclusion
  - Blood sample: hematocrit, electrolytes, serum osmolality, serum urea, serum creatinine, serum Cystatin C, serum urate, plasma renin activity (PRA), plasma aldosterone, plasma adrenaline, plasma noradrenaline, total protein, plasma NT-proBNP

### Day 1-3:

- VAS score for dyspnea
- 4-point Likert scale for edema
- Body weight and fluid balance
- o Blood pressure, heart rate, heart rhythm
- Blood sample: hematocrit, electrolytes, serum osmolality, serum urea, serum creatinine, serum Cystatin C, serum urate, PRA, plasma aldosterone, plasma adrenaline, plasma noradrenaline, total protein, plasma NT-proBNP
- Three consecutive 24h urinary collections will be performed; the first one started with the first bolus administration of loop diuretics; urinary assessment of creatinine, protein, sodium, potassium, chloride, ureum, urate, microalbuminura
- At an outpatient follow-up appointment 2-6 weeks after hospital discharge, a final blood sample with hematocrit, electrolytes, serum osmolality serum urea, serum creatinine, serum Cystatin C, serum urate and plasma NT-proBNP will be collected.
- All-cause mortality and hospital readmissions will be collected prospectively for the study cohort. The patient will receive a telephone call from a study nurse after 3, 6, 9 and 12 months

## 3.5. Study end-points

#### 3.5.1. Primary study end-point acetazolamide arm

Total urinary sodium excretion (mmol) after 24 h

## 3.5.2. Pimary study end-point for spironolactone arm

Incidence of hypo- (serum potassium <3.5mmol/L or need for oral/intravenous potassium supplements) or hyperkalemia (serum potassium >5.0mmol/L) during the entire 72 h interval after randomization.

### 3.5.3. Secondary end-points

- Relative plasma NT-proBNP change (%) after 72 h compared to admission
- Worsening renal function defined as a >0.3 mg/dL increase in serum creatinine or a
   >20% decrease in estimated glomerular filtration rate by the CKD-EPI formula
   compared to baseline at any time point before 72 h
- Persistent renal impairment, defined as persistently elevated serum creatinine levels
   >0.3 mg/dL or a >20% decrease in estimated glomerular filtration rate by the CKD-EPI formula compared to baseline at the moment of outpatient follow-up 2-6 weeks after hospital discharge.
- Peak plasma aldosterone concentration (ng/L) after 72 h
- Peak plasma renin activity (ng/mL/h) after 72 h

## 3.5.4. Other pre-specified outcome measures

- Total urinary sodium excretion (mmol) after 48 h and 72 h
- Total urine output after 24 h, 48 h and 72 h
- Change in VAS score for dyspnea at 24 h, 48 h and 72 h
- Change in 4-point Likert scale for edema at 24 h, 48 h and 72 h
- Body weight change upon hospital discharge compared to admission
- Incidence of therapy-refractory congestion defined as the need for combinational diuretic therapy with chlorthalidone, bail-out ultrafiltration or renal replacement therapy

Incidence of all-cause mortality and readmissions after 1 year

## 3.6. Statistical analysis

Continuous variables will be expressed as mean ± standard deviation when normally distributed and as median (interquartile range) in case of a non-normal distribution. Normality will be assessed by the Shapiro-Wilk The statistic. independent-samples Student's t-test and Mann-Whitney U test will be used as indicated to compare between groups. Categorical variables will be expressed as percentages and compared using Fisher's exact test or Pearson's  $\chi^2$ -test in case of a non-binary response. Statistical significance will always be set at a 2-tailed probability level of <0.05. All statistics will be performed using IBM SPSS® (Chicago, Illinois, USA) (version 22.0 for Mac).

#### 4. Potential adverse events

- Metabolic acidosis is the only agent-specific adverse event that might be expected from treatment with acetazolamide. Serum bicarbonate is monitored daily. If serum bicarbonate <22 meg/L, substitution with oral NaHCO<sub>3</sub> will be provided.
- Hyperkalemia might be expected as a potential adverse event of spironolactone, but
  this medication will be withheld when serum potassium levels are >5.0 mmol/L and
  serum potassium levels are monitored daily throughout the study.

### 5. References

1. Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB. Heart disease and stroke statistics--2013 update: A report from the

- american heart association. Circulation. 2013;127:e6-e245
- Effect of enalapril on survival in patients with reduced left ventricular ejection fractions and congestive heart failure. The solvd investigators. The New England journal of medicine. 1991;325:293-302
- 3. Cohn JN, Johnson G, Ziesche S, Cobb F, Francis G, Tristani F, Smith R, Dunkman WB, Loeb H, Wong M, et al. A comparison of enalapril with hydralazine-isosorbide dinitrate in the treatment of chronic congestive heart failure. *N Engl J Med*. 1991;325:303-310
- Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH.
   The effect of carvedilol on morbidity and mortality in patients with chronic heart failure.
   U.S. Carvedilol heart failure study group. N Engl J Med. 1996;334:1349-1355
- 5. The cardiac insufficiency bisoprolol study ii (cibis-ii): A randomised trial. *Lancet*. 1999;353:9-13
- 6. Effect of metoprolol cr/xl in chronic heart failure: Metoprolol cr/xl randomised intervention trial in congestive heart failure (merit-hf). *Lancet*. 1999;353:2001-2007
- Packer M, Coats AJ, Fowler MB, Katus HA, Krum H, Mohacsi P, Rouleau JL, Tendera M, Castaigne A, Roecker EB, Schultz MK, DeMets DL. Effect of carvedilol on survival in severe chronic heart failure. N Engl J Med. 2001;344:1651-1658
- 8. Flather MD, Shibata MC, Coats AJ, Van Veldhuisen DJ, Parkhomenko A, Borbola J, Cohen-Solal A, Dumitrascu D, Ferrari R, Lechat P, Soler-Soler J, Tavazzi L, Spinarova L, Toman J, Bohm M, Anker SD, Thompson SG, Poole-Wilson PA. Randomized trial to determine the effect of nebivolol on mortality and cardiovascular hospital admission in elderly patients with heart failure (seniors). Eur Heart J. 2005;26:215-225
- 9. Cohn JN, Tognoni G. A randomized trial of the angiotensin-receptor blocker valsartan in chronic heart failure. *N Engl J Med*. 2001;345:1667-1675
- 10. Pfeffer MA, Swedberg K, Granger CB, Held P, McMurray JJ, Michelson EL, Olofsson B, Ostergren J, Yusuf S, Pocock S, Investigators C, Committees. Effects of candesartan on mortality and morbidity in patients with chronic heart failure: The charm-overall

- programme. Lancet. 2003;362:759-766
- 11. Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized aldactone evaluation study investigators. N Engl J Med. 1999;341:709-717
- 12. Zannad F, McMurray JJ, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pocock SJ, Pitt B. Eplerenone in patients with systolic heart failure and mild symptoms. N Engl J Med. 2011;364:11-21
- 13. Swedberg K, Komajda M, Bohm M, Borer JS, Ford I, Dubost-Brama A, Lerebours G, Tavazzi L, Investigators S. Ivabradine and outcomes in chronic heart failure (shift): A randomised placebo-controlled study. *Lancet*. 2010;376:875-885
- 14. Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004;350:2140-2150
- 15. Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L.
  The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl
  J Med. 2005;352:1539-1549
- 16. Moss AJ, Hall WJ, Cannom DS, Klein H, Brown MW, Daubert JP, Estes NA, 3rd, Foster E, Greenberg H, Higgins SL, Pfeffer MA, Solomon SD, Wilber D, Zareba W. Cardiac-resynchronization therapy for the prevention of heart-failure events. N Engl J Med. 2009;361:1329-1338
- 17. Tang AS, Wells GA, Talajic M, Arnold MO, Sheldon R, Connolly S, Hohnloser SH, Nichol G, Birnie DH, Sapp JL, Yee R, Healey JS, Rouleau JL. Cardiac-resynchronization therapy for mild-to-moderate heart failure. N Engl J Med. 2010;363:2385-2395
- 18. Adams KF, Jr., Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP. Characteristics and outcomes of patients hospitalized for heart failure in the united states: Rationale, design, and preliminary

- observations from the first 100,000 cases in the acute decompensated heart failure national registry (adhere). *Am Heart J.* 2005;149:209-216
- 19. Forman DE, Butler J, Wang Y, Abraham WT, O'Connor CM, Gottlieb SS, Loh E, Massie BM, Rich MW, Stevenson LW, Young JB, Krumholz HM. Incidence, predictors at admission, and impact of worsening renal function among patients hospitalized with heart failure. J Am Coll Cardiol. 2004;43:61-67
- 20. Testani JM, Chen J, McCauley BD, Kimmel SE, Shannon RP. Potential effects of aggressive decongestion during the treatment of decompensated heart failure on renal function and survival. *Circulation*. 2010;122:265-272
- 21. Testani JM, Cappola TP, Brensinger CM, Shannon RP, Kimmel SE. Interaction between loop diuretic-associated mortality and blood urea nitrogen concentration in chronic heart failure. *J Am Coll Cardiol*. 2011;58:375-382
- 22. Testani JM, Kimmel SE, Dries DL, Coca SG. Prognostic importance of early worsening renal function after initiation of angiotensin-converting enzyme inhibitor therapy in patients with cardiac dysfunction. *Circ Heart Fail*. 2011;4:685-691
- 23. Metra M, Davison B, Bettari L, Sun H, Edwards C, Lazzarini V, Piovanelli B, Carubelli V, Bugatti S, Lombardi C, Cotter G, Dei Cas L. Is worsening renal function an ominous prognostic sign in patients with acute heart failure? The role of congestion and its interaction with renal function. *Circulation. Heart failure*. 2012;5:54-62
- 24. Felker GM, Lee KL, Bull DA, Redfield MM, Stevenson LW, Goldsmith SR, LeWinter MM, Deswal A, Rouleau JL, Ofili EO, Anstrom KJ, Hernandez AF, McNulty SE, Velazquez EJ, Kfoury AG, Chen HH, Givertz MM, Semigran MJ, Bart BA, Mascette AM, Braunwald E, O'Connor CM. Diuretic strategies in patients with acute decompensated heart failure. *N Engl J Med*. 2011;364:797-805
- 25. Schnermann J. Juxtaglomerular cell complex in the regulation of renal salt excretion. *Am J Physiol*. 1998;274:R263-279
- 26. Knauf H, Mutschler E. Sequential nephron blockade breaks resistance to diuretics in

edematous states. Journal of cardiovascular pharmacology. 1997;29:367-372

27. Cleland JG, Dargie HJ, Ford I. Mortality in heart failure: Clinical variables of prognostic value. *Br Heart J.* 1987;58:572-582